CLINICAL TRIAL: NCT00003348
Title: Phase I Trial of BCNU Plus O6-Benzylguanine in the Treatment of Patients With Recurrent, Persistent or Progressive Cerebral Anaplastic Gliomas
Brief Title: Carmustine Plus O(6)-Benzylguanine in Treating Patients With Recurrent or Progressive Gliomas of the Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066327; DUMC-1094-99-6R5; DUMC-929-97-6R3; DUMC-980-98-6R4; NCI-T94-0080
Record Dates: First submitted 1999-11-01; First posted 2004-08-16 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — O(6)-benzylguanine; Carmustine

INTERVENTIONS:
Drug: O6-benzylguanine
Drug: carmustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of carmustine plus O(6)-benzylguanine in treating patients who have recurrent or progressive gliomas of the brain.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of carmustine when administered following O6-benzylguanine in patients with recurrent, persistent, or progressive cerebral anaplastic gliomas. II. Characterize the toxic effects associated with this treatment regimen in these patients. III. Observe patients for clinical antitumor response when treated with this regimen.

OUTLINE: Patients are stratified according to prior nitrosourea administration (yes or no). (Prior nitrosoureas stratum closed) An initial cohort of 3 patients per stratum is treated with intravenous O6-benzylguanine followed approximately 1 hour later by intravenous carmustine every 6 weeks. Additional cohorts of 3-6 patients are treated with escalating doses of carmustine until dose limiting toxicity (DLT) is observed. The maximum tolerated dose is defined as the dose at which no more than 1 of 6 patients experiences DLT. Courses are repeated every 6 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 24-56 patients (12-28 per stratum) will be accrued in 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent, persistent, or progressive glioblastoma multiforme or anaplastic astrocytoma diagnosed by biopsy/resection Evaluable residual disease by MRI or CT scan

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: SGOT no greater than 2.5 times upper limit of normal Bilirubin within normal limits Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min BUN no greater than 25 mg/dL Pulmonary: DLCO greater than 80% predicted Other: Not pregnant or nursing Fertile patients must use effective contraceptive method during and for 2 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks since prior nitrosourea, procarbazine, or mitomycin) and recovered Endocrine therapy: Concurrent corticosteroid therapy must be stable for at least 1 week prior to study, if clinically possible Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 1998-05; Primary Completion 2000-08 (Actual); Study Completion 2000-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States